CLINICAL TRIAL: NCT01778465
Title: Effect of Low Dietary Salicylate on Biochemical Markers of Aspirin Exacerbated Respiratory Disease
Brief Title: Effect of Dietary Salicylate in Aspirin Exacerbated Respiratory Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 103330
Record Dates: First submitted 2013-01-26; First posted 2013-01-29 (Estimated); Results first posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2015-03

CONDITIONS: Chronic Rhinosinusitis; Aspirin Exacerbated Respiratory Disease; Asthma; Aspirin Sensitivity
Keywords: Chronic Rhinosinusitis; Aspirin exacerbated respiratory disease; Asthma; Aspirin sensitivity; Salicylate
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low salicylate diet, then Normal Diet (Experimental): Patients followed a low salicylate diet for one week, then they followed a Normal diet for another week.
  Interventions: Behavioral: Low salicylate diet
- Normal diet, then Low Salicylate diet (Experimental): Patients followed a Normal diet for one week, then they followed a Low Salicylate diet for another week.
  Interventions: Behavioral: Normal Diet

INTERVENTIONS:
Behavioral: Low salicylate diet — Participants followed a 7 days period under a Low salicylate diet
  Other Names: Dietary salicylate
  Arms: Low salicylate diet, then Normal Diet
Behavioral: Normal Diet — Participants followed a 7 days period under a Normal Diet
  Arms: Normal diet, then Low Salicylate diet

SUMMARY:
Aspirin-Exacerbated Respiratory Disease, or AERD, consists of aspirin sensitivity, asthma and nasal polyps. It is currently managed by chronic steroid use, multiple endoscopic sinus surgeries and/or aspirin desensitization. However, these treatments have potential adverse effects.

A theory has been postulated that decreasing the level of dietary salicylates may help in long-term control of disease. A current trial is in the works to evaluate the clinical outcomes of decreased salicylate, but measurements of biochemical markers of disease has not yet been done. The hypothesis is that decreased dietary salicylates will result in a decrease in urinary salicylates and inflammatory markers of disease, cys-leukotrienes, which are typically elevated in this disease.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* Aspirin-exacerbated respiratory disease

Exclusion Criteria:

* recent use of Prednisone or other systemic steroids (greater than 3 doses in past 3 months)
* Endoscopic sinus surgery or polypectomy within the past 6 months
* Other significant systemic disease, including renal failure, or immunocompromised state.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-05; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leigh J Sowerby, MD, Principal Investigator — Lawson HRI
Locations (1):
- St. Joseph's Health Care, London, Ontario, Canada

REFERENCES:
- [Derived] Sowerby LJ, Patel KB, Schmerk C, Rotenberg BW, Rocha T, Sommer DD. Effect of low salicylate diet on clinical and inflammatory markers in patients with aspirin exacerbated respiratory disease - a randomized crossover trial. J Otolaryngol Head Neck Surg. 2021 Apr 23;50(1):27. doi: 10.1186/s40463-021-00502-4. PMID 33892819

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Salicylate Diet, Then Normal Diet: Participants followed a low salicylate diet for 7 days, then they started a period of 7 days on Normal diet.
- Normal Diet, Then Low Salicylate Diet: Participants followed a normal diet for 7 days, then they started a period of 7 days on Low Salicylate Diet
Period: First Intervention (7 Days)
Arm/Group | Low Salicylate Diet, Then Normal Diet | Normal Diet, Then Low Salicylate Diet
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0
Period: Second Intervention (7 Days)
Arm/Group | Low Salicylate Diet, Then Normal Diet | Normal Diet, Then Low Salicylate Diet
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants followed a low salicylate diet for one week. Then, participants continued with a normal diet for one week.
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Urinary Levels of Cys-Leukotrienes
Time Frame: 14 days after commencement
Measure: Median (Inter-Quartile Range); unit: pg/ml
Groups:
- Low Salicylate Diet: Patients followed a low salicylate diet for one week
- Normal Diet: Patients followed a Normal diet for one week.
Arm/Group | Low Salicylate Diet | Normal Diet
Number analyzed (Participants) | 7 | 7
pg/ml | 874.05 [182.60 to 1404.01] | 771.99 [651.23 to 1979.22]

2. Primary Outcome: Urinary Salicyluric Acid Levels
Time Frame: 14 days after commencement
Measure: Median (Inter-Quartile Range); unit: ng/ml
Groups:
- Normal Diet: Participants followed a normal diet for 7 days
Arm/Group | Low Salicylate Diet | Normal Diet
Number analyzed (Participants) | 7 | 7
ng/ml | 44.21 [20.23 to 54.9] | 23.82 [15.7 to 70.08]

3. Primary Outcome: Urinary Salicylic Acid Levels
Time Frame: 14 days after enrollment
Measure: Median (Inter-Quartile Range); unit: ng/ml
Groups:
- Low Salicylate Diet: Participants followed a low salicylate diet for 7 days
Arm/Group | Low Salicylate Diet | Normal Diet
Number analyzed (Participants) | 7 | 7
ng/ml | 0.6 [0.46 to 3.88] | 0.92 [0.4 to 1.2]

4. Primary Outcome: Urinary Creatinine Levels
Time Frame: 14 days after commencement
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Low Salicylate Diet | Normal Diet
Number analyzed (Participants) | 7 | 7
mmol/L | 9.9 [3.7 to 15] | 15.3 [6.2 to 18.8]

5. Secondary Outcome: Sino-Nasal Outcome Test (SNOT-22)
Description: The Sino-Nasal Outcome Test (SNOT-22) is a validated 22-item Chronic rhinosinusitis-specific instrument which is scored using a scale where 0="No problem", 1="Very mild problem", 2="Mild or slight problem", 3="Moderate problem", 4="Severe problem", and 5="Problem as bad as it can be". Higher scores on the SNOT-22 survey items suggest worse patient functioning or symptom severity (total score range: 0-110)
Time Frame: 14 days after commencement
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Low Salicylate Diet | Normal Diet
Number analyzed (Participants) | 7 | 7
score on a scale | 44 [22 to 53] | 66 [43 to 83]

ADVERSE EVENTS:
Arm/Group | Low Salicylate Diet | Normal Diet
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No